CLINICAL TRIAL: NCT02494037
Title: The Canadian/US Integrative Oncology Study (CUSIOS): Advanced Integrative Oncology Treatment for Patients With Advanced Stage Cancer: A Prospective Outcomes Study
Brief Title: The Canadian/US Integrative Oncology Study
Acronym: CUSIOS
Status: Completed | Type: Observational
Sponsor: The Canadian College of Naturopathic Medicine (Other)
Collaborators: Bastyr University (Other); Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 3974
Record Dates: First submitted 2015-07-03; First posted 2015-07-10 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study describes the survival outcomes of advanced stage breast, colorectal, ovarian and pancreatic cancer patients receiving advanced integrative oncology (AIO) treatment at participating North American integrative oncology clinics. This study also aims to describe the integrative treatments recommended by naturopathic doctors (NDs) for these participants alongside their conventional care treatments. Sub-studies will evaluate health-related quality of life, cost of cancer care, and qualitative experience of care in a subset of Canadian participants.

DETAILED DESCRIPTION:
It is estimated that between 50 and 80% of cancer patients in the United States (US) supplement their conventional oncology treatment regimen with some form of complementary or alternative medicine therapy or practice. A smaller percentage of these patients receive care from naturopathic doctors (NDs) who are board certified in naturopathic oncology (Fellows of the American Board of Naturopathic Oncology, FABNO) or have equivalent experience in caring for cancer patients and from traditional Chinese medicine (TCM) providers with advanced training in oncology (DAOM or physicians with training in TCM). This level of care is being defined here as advanced integrative oncology (AIO). AIO clinics provide comprehensive science- and experience-based naturopathic and Chinese medical oncology integrated with each patient's conventional medical treatment.

Although there have been some studies of complementary and alternative medicine use by cancer patients, little is known about the effectiveness of the naturopathic medicine and TCM provided to people with cancer in an integrative setting. While there is scientific evidence supporting specific treatments that are commonly used, systematic study of their effectiveness (especially when used in combination as commonly recommended) is virtually non-existent. An early step in the evaluation of clinical outcomes associated with AIO is to take a health service approach and seek to answer the question: "Does exposure to AIO services improve the clinical outcomes of patients with advanced stage cancer?"

The survival outcome of advanced stage breast, colorectal, pancreatic, and ovarian cancer patients treated at multiple naturopathic oncology clinics in North America will be tracked and compared to outcomes from the SEER (Surveillance, Epidemiology and End Results) database in order to address the fundamentally important question of whether or not AIO has a beneficial impact on survival. Involvement of a total of twelve clinics from Canada and the US will allow the recruitment of a sufficient sample size to address this question as well as provide outcomes that enhance the generalizability for AIO across North America.

ELIGIBILITY:
Inclusion Criteria:

* A new patient coming in for a first office call (FOC) with a participating site investigator for their cancer or a current patient whose FOC with a participating investigator for their cancer was after study start date of January 1, 2015
* ≥18 years of age
* Able to understand study design and provide signed informed consent to enrollment
* Confirmed diagnosis of one of the following cancers: stage 4/metastatic breast, stage 4/metastatic colorectal, stage 3 or 4/metasatic ovarian, or stage 3 or 4/metastatic pancreatic
* Canadian participants with a visit <3 months post-FOC are eligible for the HRQOL sub-study
* Participants must be governed by the laws of the country within which they are receiving AIO care

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stage 4 or metastatic breast or colorectal cancer patients and all stage 3 or 4 or metastatic ovarian and pancreatic cancer patients seeking care at the participating AIO clinical sites meeting inclusion/exclusion criteria are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Survival | From date of diagnosis of stage IV or metastatic disease to 3 years post enrollment
  To measure the survival of AIO-treated patients as compared to survival data from the SEER database

SECONDARY OUTCOMES:
Description of Integrative care | At enrollment and up to 3 years
  AIO treatment recommendations for cancer and conventional oncology treatment data will be collected to describe the cancer treatments recommended and/or used by cancer patients across the treatment cohort. AIO treatment recommendations will be abstracted from AIO chart notes for all study participants for the first AIO clinic visit and up to 3 years. Concurrent conventional oncology treatment data will also be abstracted from conventional oncology medical charts.
Health-Related Quality of Life (HRQOL) | At baseline and 3 and 6 months and 1, 2 and 3 years thereafter.
  Self-reported HRQOL data will be collected from a subgroup of Canadian AIO-treated patients who had at least two AIO visits within three months of first AIO clinic visit using validated questionnaires commonly used in integrative oncology research settings. Instruments to be used in the HRQOL assessment include the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) to measure general health status and function, Measure Yourself Concerns and Wellbeing (MYCaW) to identify cancer-related concerns, and Edmonton Symptom Assessment Scale (ESAS) to assess common cancer symptoms.
Cost of Cancer Care | At baseline and 6 months, 1 year, 2 years, and 3 years thereafter
  A sub group of Canadian AIO-treated patients will be enrolled to estimate direct healthcare, direct non-healthcare, and indirect non-healthcare costs from a societal perspective. This includes costs incurred by the healthcare payer (i.e. government or private insurers), the patient/family (i.e. co-payment or full payment for medicines and/or care) and by the society at large (i.e. costs of reduced productivity). Patients will self-report these costs using questionnaires developed by the research team in collaboration with a health economist.
Qualitative Experience of Care (QEC) | At baseline and 3 months, 6 months, 1 year, 2 years, and 3 years thereafter.
  A Sub group of Canadian AIO-treated patients and NDs at each Canadian clinic will be enrolled to understand the benefits and challenges of AIO care from a qualitative perspective. Through interviews conducted by a qualitative researcher, we will help to more fully understand the experiences of study participants and the subjective impact of naturopathic interventions both from the perspective of the study participants themselves and from the perspective of their ND.

CONTACTS AND LOCATIONS:
Overall Officials: Dugald Seely, ND, MSc, Principal Investigator — Canadian College of Naturopathic Medicine; Leanna Standish, ND, PhD, FABNO, Principal Investigator — Bastyr University
Locations (12):
- United States (7):
  - Naturopathic Specialists, LLC (NSL), Scottsdale, Arizona
  - Hawaii Integrative Oncology, Lokahi Health Center, Inc. (LHC), Kailua, Hawaii
  - Salish Cancer Center (SCC), Fife, Washington
  - Seattle Integrative Cancer Center, Seattle, Washington
  - Advanced Integrative Medical Science (AIMS) Institute, Seattle, Washington
  - Bastyr Center for Natural Health, Seattle, Washington
  - Tree of Health Integrative Medicine, Woodinville, Washington
- Canada (5):
  - Integrated Health Clinic Cancer Care Centre, Fort Langley, British Columbia
  - Vital Victoria Naturopathic Clinic Ltd., Victoria, British Columbia
  - HealthSource Integrative Medical Centre, Kitchener, Ontario
  - Ottawa Integrative Cancer Centre (OICC), Ottawa, Ontario
  - Marsden Centre for Excellence in Integrative Medicine, Vaughan, Ontario